CLINICAL TRIAL: NCT01203007
Title: A Pilot Study of 6 Months Diet Intervention in Food Sensitive Patients With IgA Nephropathy
Brief Title: Diet Intervention in Food Sensitive Patients With IgA Nephropathy
Acronym: DIIGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: University Hospital, Linkoeping (Other); Haukeland University Hospital (Other); Smerud Medical Research International AS (Other)
Responsible Party: Bengt Fellström, Uppsala University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMR-2259
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: IGA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored diet (Experimental): Tailored diet according to demonstrated food sensitivity
  Interventions: Dietary Supplement: Tailored diet
- Low-antigen content (LAC) diet (Experimental): Low-antigen content diet
  Interventions: Dietary Supplement: Low antigen content diet

INTERVENTIONS:
Dietary Supplement: Tailored diet — Tailored diet according to demonstrated food sensitivity, 6 months
  Arms: Tailored diet
Dietary Supplement: Low antigen content diet — Low-antigen content diet for one month
  Arms: Low-antigen content (LAC) diet

SUMMARY:
The purpose of this study is to assess whether a tailored diet, eliminating antigens to which IgA nephropathy patients have demonstrated sensitivity, will have an effect on proteinuria, renal function and other immunological variables.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years
* IgA nephropathy (IgAN), verified by biopsy
* Proteinuria > 1 g/24 h
* Having signed informed consent form

Exclusion Criteria:

* Participation in another clinical trial
* Patients with celiac disease
* Introduction of an angiotensin-converting enzyme (ACE) inhibitor or angiotensin II receptor blockers (ARB) during the last three months prior to inclusion
* Patients treated with immunosuppressive or systemic corticosteroid drugs within the last twelve months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Proteinuria | 6 months

SECONDARY OUTCOMES:
Renal function | 6 months
  Glomerular filtration rate (GFR)
IgA/IgG immune complexes, incl. glycosylation | 6 months
IgA/IgG to dietary antigens | 6 months
Hematuria | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hilde K Smerud, MScPharm, Study Director — Uppsala University Hospital
Locations (3):
- Haukeland University Hospital, Bergen, Norway
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Uppsala University Hospital, Uppsala